CLINICAL TRIAL: NCT04715347
Title: Interstitial Lung Disease Within a Lung Cancer Screening
Acronym: ILD
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017TC011
Record Dates: First submitted 2020-07-27; First posted 2021-01-20 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interstitial lung disease is a devastating lung condition with terrible outcomes. Lung cancer is the world's leading cause of cancer related death. Unlike breast and bowel cancer, there is no lung cancer screening programme in the UK. However, there are a number of pilot lung cancer screening programmes taking place including one in Manchester. The CT scans used in lung cancer screening programmes pick up other lung conditions out with lung cancer, including interstitial lung disease. This provides a unique opportunity to diagnose interstitial lung disease at an early and non-symptomatic stage where treatment can be initiated early to halt progression of disease and development of symptoms. The investigators aim to determine how much (prevalence) interstitial lung disease can be picked up in a lung cancer screening programme and how these cases would compare to those diagnosed with interstitial lung disease through the 'standard' way in the clinics.

The investigators hypothesis that the patients diagnosed through the screening programmes will have an earlier stage of disease with less symptoms. If this is to be the case, this would provide researchers with the opportunity to diagnose interstitial lung disease through lung cancer screening programmes and initiate treatment early.

DETAILED DESCRIPTION:
The Manchester Early Detection of Lung Disease Pilot (lung cancer screening programme) is already under way and has been for the past 12 months. A total of 1,384 individuals had a CT scan as part of this service. From these, several individuals (around 40) have been diagnosed with likely interstitial lung disease (ILD) and been referred to the regional ILD clinic at the University Hospital of South Manchester (UHSM; Wythenshawe). These patients are due to attend the clinic soon.

Individuals attending the regional ILD clinic as a 'new referral' will be invited to participate. Inclusion and exclusion criteria will be evaluated, and suitable participants will be provided with a patient information sheet (PIS) on the same day prior to written consent being obtained for enrolment into the study. Individuals will be given as much time as needed to read the PIS and ask relevant questions. We will recruit patients from two groups:

* Group 1: ILD diagnosed through the Manchester Early Detection of Lung Disease Pilot (lung cancer screening programme) and
* Group 2: age and sex matched individuals with ILD diagnosed through standard non-screening pathway

Participants will be asked to fill out a number of health-related questionnaires in addition to the standard care they will receive as part of their clinic visit. No extra tests will be performed as a result of this study, the only additional information required is related to the questionnaires. These questionnaires will focus on quality of life and symptom burden and will on average take 10-15 minutes to complete. The information gathered from their clinic visit (including any tests performed) will also be collected and used for research purposes. Once complete, the results between group 1 and group 2 will be compared.

Overall there will be three time points in the study for each participant to fill out questionnaires. This will be at the baseline visit (as above) and also at 6 months and 12 months. The 6 month and 12 month questionnaires will be completed by participants, with as required help from the research team, at a follow-up clinic visit if one is set up (ILD clinic patients are often seen back in clinic at these time points). If not clinic appointment is set up at these time points, the questionnaires will be posted to the participants for self-completion at home with help offered over the phone as required.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Ever-smoker
* MDT diagnosis of ILD that has been detected through lung cancer screening or standard non-screening pathway
* Attended the regional ILD clinic

Exclusion Criteria:

* Unable to complete self-report questionnaire measures
* Unable to provide written informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals attending the regional ILD clinic as a 'new referral' who have been referred from a lung cancer screening programme or through a standard non-screening pathway will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of ILD in participants of a community-based lung cancer screening programme. | 2 years 6 months
  This will be determined through analysing the prevalence of ILD in participants of the MCIP lung cancer screening pilot programme

SECONDARY OUTCOMES:
Comparison of the symptom and psychological burden at diagnosis between patients diagnosed through a screening programme and patients diagnosed through routine care | 2 years
  This will be determined through standardised clinical history pro forma's
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using VAS questionnaires | through study completion, an average of 2 years
  Using VAS questionnaires with a scale of the worst to none
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using FSS questionnaire | through study completion, an average of 2 years
  Using FSS questionnaire with a scale of 1-7. With 1 being strong disagreement and 7 being strong agreement
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using the LCQ questionnaire | through study completion, an average of 2 years
  LCQ questionnaire with a scale of 1-7 with All the time to Never varying on the scale.
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using the UCSD-SBQ questionnaire | through study completion, an average of 2 years
  UCSD-SBQ questionnaire, which has a scale of 0-5, with 0 being none and 5 maximum
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using SF-36 questionnaire | through study completion, an average of 2 years
  Using SF-36 questionnaire.The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability
Comparison of the quality of life between patients diagnosed through a screening programme and patients diagnosed through routine care using the K-BILD questionnaire | through study completion, an average of 2 years
  K-BILD questionnaire with a scale of 1-7 , with 1 being all the time and 7 being never/ none of the time
Qualitative comparison of the radiological pattern being depicted by ATS/ERS ILD by the multidisciplinary team (MDT) agreed type between patients diagnosed through a screening programme and patients diagnosed through routine care | through study completion at Multidisiplinary Team (MDT) meetings, for an average of 2 years
  Any Interstitial lung abnormalities (ILAs) detected on screening LDCT scans were highlighted in the CT report and referred to the regional ILD MDT for review and discussion. The radiological pattern will be established from the multidisciplinary team (MDT) pro forma's, this will be a descriptive analysis.
  The MDT consists of three ILD respiratory physicians, a thoracic radiologist with an interest in ILD, two specialist ILD nurses and an MDT co-ordinator. Once discussed at the MDT, those deemed to have changes suggestive of significant ILD have been referred to the regional ILD service for assessment in the clinic.
Lung function via full pulmonary function test in patients with diagnosed ILD between patients diagnosed through a screening programme and patients diagnosed through routine care | through study completion, an average of 2 years
  Comparison of lung function averages will be determined, a full pulmonary function test (Forced vital capacity (FVC) and transfer factor (DLCO) at diagnosis). This outcome will be comparing patients who have been diagnosed through the standard non-screening pathway and the screening programme.
Lung function via shuttle walk tests (distance walked and oxygen saturation) in patients with diagnosed ILD between patients diagnosed through a screening programme and through routine care | through study completion, an average of 2 years
  Comparison of lung function averages will be determined using shuttle walk tests, distance walked and oxygen saturation (pre and immediately post test). This outcome will be comparing patients who have been diagnosed through the standard non-screening pathway and the screening programme.
Qualitative comparison of the treatment strategies between patients diagnosed with ILD through a screening programme and patients diagnosed through routine care, this is not a quantitative measure. | through study completion, an average of 2 years
  This will be assessed through the initial treatment patients received, this will be a descriptive analysis or qualitative nature .

CONTACTS AND LOCATIONS:
Overall Officials: Jill Clayton-Smith, Professor, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS foundation trust, Manchester, Greater Manchester, United Kingdom

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04715347/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT04715347/ICF_001.pdf